CLINICAL TRIAL: NCT06036771
Title: Efficacy of the Voice-activated Intelligent Personal Assistant (VIPA) Intervention on Psychosocial Well-being Among People With Parkinson's Disease: A Pilot Randomized Controlled Trial
Brief Title: Voice-activated Intelligent Personal Assistant (VIPA) Intervention for People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Angela Leung, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSEARS20221107005
Record Dates: First submitted 2023-08-21; First posted 2023-09-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2023-09

CONDITIONS: Parkinson's Disease and Parkinsonism
Keywords: sense of coherence; psychosocial well-being; Voice-activated Intelligence Personal assistant
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Intervention Model Description: 48 PWP will be randomized into the intervention group (IG) and controlled group (CG). Block randomization is performed by an independent research team member who will not be in contact with participants via a free third-party website. Allocations will only be revealed upon the commencement of the intervention period and cannot be altered.
Who Masked: Outcomes Assessor
Masking Description: outcome assessors will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voice-activated Intelligent Personal Assistant (VIPA) intervention (Experimental): IG participants will receive
  1. The developed VIPA user protocol
  2. 30-minute training session on day 1
  3. Technical support hotline
  Dosage of the intervention: PWP are encouraged to perform 10 voice commands/ day during the 8-week intervention period, self-reported usage will be documented by participants in a progress note.
  Interventions: Device: Voice-activated Intelligent Personal Assistant (VIPA)
- Usual care, no intervention provided (No Intervention): CG participants will be placed under usual care, no intervention will be provided and PWP will continue their daily life during the intervention period

INTERVENTIONS:
Device: Voice-activated Intelligent Personal Assistant (VIPA) — Apple HomePod mini is selected as the intervention medium of this study as it is the only available smart speaker that supports Cantonese
  Arms: Voice-activated Intelligent Personal Assistant (VIPA) intervention

SUMMARY:
This pilot randomized control trial (RCT) aims to develop a Voice-activated Intelligent Personal Assistance (VIPA) user protocol and study its feasibility and preliminary efficacy among 48 People with Parkinson's disease (PWP). The research questions are:

Phase 1:

1. What components should be included in the VIPA user protocol community-dwelling PWP?
2. Is it feasible to implement the VIPA intervention in the PD population?

3 focus group interviews and 3 cognitive interviews will be held to formulate the VIPA user protocol. 5 healthcare and information technology experts will be invited to rate the relevancy of the formulated protocol and the item content validity index will be calculated by the researcher.

Phase 2:

1. What is the preliminary efficacy of VIPA intervention on SOC and psychosocial well-being?
2. Can such effect sustain for 4 weeks?
3. What is the users' experience on the VIPA intervention?

48 participants will be randomized into the intervention group (IG) and control group (CG). During the 8-week intervention period, IG participants will receive the following materials:

1. User protocol
2. Designate VIPA
3. 30-minute VIPA training on day 1
4. technical support hotline. CG participants will receive usual care, no intervention will be provided to CG participants, and they will continue their daily life during the intervention period.

The researcher will compare both groups to study the feasibility and preliminary efficacy of the VIPA on the participants' psychosocial well-being and sense of coherence.

DETAILED DESCRIPTION:
Background:

Parkinson's disease (PD) is one of the two most common neurodegenerative diseases affecting millions worldwide. PD research generally focuses on motor functioning and calls for more psychosocial interventions for people with Parkinson's disease (PWP).

The proposed VIPA intervention is an artificial intelligent personal assistant commonly used within Western society but not Asian countries, facilitating users' daily living by performing audio calls, messaging, and information searching. Recent literature showed VIPA Implementation is promising for rehabilitation in older adults but warrants more interventional studies to examine its efficacy and if it applies to other illnesses. Therefore, this study will formulate a positive health-orientated VIPA intervention protocol and investigate its efficacy in promoting PWP's sense of coherence and psychosocial well-being.

Objectives of the study:

This is a 2-phase study, and the objectives are:

Phase 1:

1. To develop and validate the VIPA user protocol.
2. To examine the feasibility of the VIPA intervention.

Phase 2:

1. To investigate the preliminary efficacy of the VIPA intervention on PWP's SOC
2. To explore the users' experience of VIPA intervention among PWP.

Method:

Phase 1: 3 semi-structured focus group interviews will be held to generate items in user protocol. Another 3 cognitive interviews will be held with PWP to test the face validity and feasibility of the user protocol. 5 healthcare and information technology experts will then be invited to assess the content validity of the protocol. Any item with an item content validity index (i-CVI) score lower than 0.78 will be discarded or revised.

Phase 2: 48 participants will be randomized into the intervention group (IG) and control group (CG). During the 8-week intervention period, IG participants will receive the user protocol, a designated VIPA, a 30-minute VIPA training on day 1, and technical support hotline. CG participants will receive usual care (no intervention will be provided to CG participants), and they will continue their daily life during the intervention period. The 13-item Sense of Coherence Scale (SOC-13) will be set as the primary outcome, and secondary outcomes are: 1. University of California, Los Angeles (UCLA) three-item loneliness scale; 2. Parkinson's Disease Questionnaire (PDQ-8); 3. EuroQol-5 dimension-5 level; 4. Mental Health Continuum Short Form; 5. System Usability Scale; 6. Brief Resilient Coping Scale; 7. Montreal Cognitive Assessment; and 8. Self-report VIPA usage.

12 participants will then be selected through extreme case sampling to partake in explanatory, in-depth interviews based on their SOC-13 score differences between baseline and post-intervention tests to explore VIPA user experience.

Data analysis:

For qualitative data, content analysis will be used in phase 1, while in phase 2, in-depth interview data will be analyzed through deductive thematic analysis according to the salutogenic model. Quantitative data, such as demographic data, will be presented with descriptive statistics. Chi-square test and independent t-test will be performed for baseline comparison. Generalized Estimating Equations will be used to analyze group differences in all primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese-speaking Hong Kong permanent resident
* Diagnosed with Parkinson's disease
* Level 1-4 in the H&Y scale (Hoehn & Yahr, 1967)
* Not currently using or owning VIPA
* Has stable Wi-Fi connection at home.

Exclusion Criteria:

* PWP or their caregivers that fails to provide valid consent
* Individuals with hearing loss in both ears
* Severe voice impairment
* Dementia patients (MoCA score <21)
* PWP will leave Hong Kong during the intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-08-06 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
13-item Sense of Coherence Scale | [Time Frame: Baseline; 8 weeks; 12 weeks]
  The 13-item Sense of Coherence Scale is a 13 item, 7-point Likert scale that measures PWP's sense of coherence. Its score ranges from 13-91, with a higher score representing a higher sense of coherence.

SECONDARY OUTCOMES:
UCLA three-item loneliness scale | [Time Frame: Baseline; 8 weeks; 12 weeks]
  The UCLA three-item loneliness scale is a 3 item, 3-point Likert scale that measures PWP's perceived loneliness. Its score ranges from 3-9, with a higher score indicating a more lonely sensation.
Parkinson's Disease Questionnaire (PDQ-8) | [Time Frame: Baseline; 8 weeks; 12 weeks]
  Parkinson's Disease Questionnaire (PDQ-8) is an 8 item, 5-point Likert scale commonly adopted to measure PWP's quality of life. The higher summative score indicates a lower quality of life experienced.
EuroQol- 5 dimension- 5 level | [Time Frame: Baseline]
  EuroQol- 5 dimension- 5 level utilized a visual analogue scale from 1-100 and 5 descriptive statements to explore an individual's quality of life. This scale is adopted to validate the newly translated PDQ-8
Mental Health Continuum Short Form | [Time Frame: Baseline; 8 weeks; 12 weeks]
  The Mental Health Continuum Short Form is a 14 item, 6-point Likert scale measuring PWP's psychosocial well-being. Its score ranges from 0-70, with a higher score indicating higher psychosocial well-being.
Brief Resilient Coping Scale | [Time Frame: Baseline; 8 weeks; 12 weeks]
  The Brief Resilient Coping Scale is a 4 item, 5-point Likert scale measuring an individual's coping. Its score ranges from 4-20, with a higher score indicating better coping.
Montreal Cognitive Assessment (MoCA) | [Time Frame: Screening]
  The Montreal Cognitive Assessment (MoCA) is a professional administrated assessment to evaluate an individual's cognitive functioning. This scale will be first administered to screen out PWP with dementia. Its score ranges from 0-30, with a higher score representing higher cognitive functioning.
System Usability Scale | [Time Frame: 8 weeks]
  System Usability Scale is a 10 item,5-point Likert scale that assess the usability of the implemented intervention. Its score ranges from 0-100, with a higher score indicates a higher usability
Self-report VIPA usage | [Time Frame: 8 weeks]
  PWP will report self-report VIPA usage across the intervention period. A logbook will be provided to PWP to log down their daily usage.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold A, Kolody S, Comeau A, Miguel Cruz A. What does the literature say about the use of personal voice assistants in older adults? A scoping review. Disabil Rehabil Assist Technol. 2024 Jan;19(1):100-111. doi: 10.1080/17483107.2022.2065369. Epub 2022 Apr 22. PMID 35459429
- [Background] Antonovsky, A. (1987). Unravelling the mystery of health: How people manage stress
- [Background] Jenkinson, C., Fitzpatrick, R., Peto, V., Greenhall, R., & Hyman, N. (1997). The PDQ-8: development and validation of a short-form Parkinson's disease questionnaire. Psychology and Health, 12(6), 805-814.
- [Background] Szende A, Janssen B, Cabases J, editors. Self-Reported Population Health: An International Perspective based on EQ-5D [Internet]. Dordrecht (NL): Springer; 2014. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK500356/ PMID 29787044
- [Background] Lamers SM, Westerhof GJ, Bohlmeijer ET, ten Klooster PM, Keyes CL. Evaluating the psychometric properties of the Mental Health Continuum-Short Form (MHC-SF). J Clin Psychol. 2011 Jan;67(1):99-110. doi: 10.1002/jclp.20741. PMID 20973032
- [Background] Brooke, J. (1996). SUS-A quick and dirty usability scale. Usability evaluation in industry, 189(194), 4-7.
- [Background] Sinclair VG, Wallston KA. The development and psychometric evaluation of the Brief Resilient Coping Scale. Assessment. 2004 Mar;11(1):94-101. doi: 10.1177/1073191103258144. PMID 14994958
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Reggiani P, Gridelli B, Colledan M, Rossi G, Lucianetti A, Galmarini D, Fassati LR. Rescue FK506 early conversion for refractory rejection after pediatric liver transplantation: experience in 20 children. Transpl Int. 1998;11 Suppl 1:S272-4. doi: 10.1007/s001470050477. PMID 9664995
- [Background] Cools CI, de Vries NM, Bloem BR. Happiness: A Novel Outcome in Parkinson Studies? J Parkinsons Dis. 2020;10(3):1261-1266. doi: 10.3233/JPD-201999. PMID 32568107
- [Background] NIEHS(2021). Neurodegenerative Diseases. Retrieved from United States Department of Health and Human Services, The National Institute of Environmental Health Sciences (NIEHS) Web site: https://www.niehs.nih.gov/research/supported/health/neurodegenerative/index.cfm